CLINICAL TRIAL: NCT00002055
Title: A Double-Blind Group Comparative Study To Evaluate the Long-Term Safety and Effectiveness of Two Different Doses of Aerosol Pentamidine in the Prophylaxis of Pneumocystis Carinii Pneumonia in AIDS Patients With Multiple Episodes of PCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisons (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 022D; 88-7
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-01

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Pentamidine; Dose-Response Relationship, Drug; Aerosols; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Pentamidine

INTERVENTIONS:
Drug: Pentamidine isethionate

SUMMARY:
To evaluate and compare the safety, tolerability, and effectiveness of long-term biweekly administration of 1 of 2 doses of aerosol pentamidine when used as a prophylactic agent in patients who have had multiple episodes of AIDS associated Pneumocystis carinii pneumonia (PCP).

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine (AZT).

Patients must have:

* AIDS.
* Recovered from their most recent episode of Pneumocystis carinii pneumonia (PCP). Patients must be at least 2 weeks status post therapy for acute PCP.
* Adequate pulmonary function (vital capacity = or > 65 percent of predicted; forced expiratory volume, 1 s = or > 55 percent of total FEV; and corrected pulmonary diffusion capacity > 50 percent of predicted).
* Patients must be free of acute medical problems.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* AIDS-defining opportunistic infection prior to entry such as toxoplasmosis and cryptococcosis.
* Pulmonary Kaposi's sarcoma.
* Asthma poorly controlled by medication.
* Receiving active therapy for tuberculosis.

Concurrent Medication:

Excluded:

* Active therapy for tuberculosis.

Patients with the following are excluded:

* Requiring ongoing active therapy for an opportunistic infection at time of study entry.
* AIDS-defining opportunistic infection prior to study entry such as toxoplasmosis and cryptococcosis.
* Pulmonary Kaposi's sarcoma.
* Unwilling to sign informed consent.
* Asthma poorly controlled by medication.
* Unwilling to cooperate with study procedures.
* Receiving active therapy for tuberculosis.

Prior Medication:

Excluded within 30 days of study entry:

* Antiretrovirals (other than zidovudine (AZT)).
* Immunomodulating agents.
* Corticosteroids.

Prior Treatment:

Excluded within 7 days of study entry:

* Transfusion.
* Patient cannot be transfusion dependent (requiring blood transfusion more than once per month).

Active substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Georgetown Univ, Washington D.C., District of Columbia
  - Veterans Administration Med Ctr, Washington D.C., District of Columbia
  - Northwestern Univ Med School, Chicago, Illinois
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts

REFERENCES:
- [Background] Lavelle J, Murphy R, Harding P, Pierce P. Aerosolized pentamidine prophylaxis following Pneumocystis carinii pneumonia in patients with AIDS. Int Conf AIDS. 1990 Jun 20-23;6(2):374 (abstract no 2083)
- [Background] Murphy RL, Lavelle JP, Allan JD, Gordin FM, Dupliss R, Boswell SL, Waskin HA, Davies SF, Graziano FM, Saag MS, et al. Aerosol pentamidine prophylaxis following Pneumocystis carinii pneumonia in AIDS patients: results of a blinded dose-comparison study using an ultrasonic nebulizer. Am J Med. 1991 Apr;90(4):418-26. PMID 2012082